CLINICAL TRIAL: NCT02208336
Title: Evaluation of a Data Driven System for Insuring Timely Monitoring for Brain Tumor Patients for Management of Myelosuppression
Brief Title: Electronic Medical Record Review in Monitoring the Effects of Adherence on Myelosuppression and Morbidity in Patients With Newly Diagnosed Brain Tumors Receiving Temozolomide and Radiation Therapy
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CCCWFU 99210; NCI-2014-01602 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 99210 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2014-08-01; First posted 2014-08-05 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (electronic medical record review): Patients' electronic medical records are reviewed for adherence, severe myelosuppression, and patient morbidity retrospectively and prospectively.
  Interventions: Other: medical chart review

INTERVENTIONS:
Other: medical chart review — Ancillary studies
  Other Names: chart review

SUMMARY:
This research trial studies electronic medical record review in monitoring the effects of adherence on myelosuppression and morbidity in patients with newly diagnosed brain tumors receiving temozolomide and radiation therapy. Myelosuppression is a condition in which bone marrow activity is decreased, resulting in fewer red blood cells, white blood cells, and platelets and is a side effect of some cancer treatments. Morbidity is a term that refers to having a symptom of disease or medical problems caused by a treatment. Monitoring patients' electronic medical records to compare side effects, such as myelosuppression and morbidity, with treatment adherence may be a way to enhance patient care by organizing data for medical staff.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Retrospectively measure the frequency of nonadherence with established monitoring guidelines in the target patient population.

II. Retrospectively assess the impact of nonadherence events on myelosuppression severity and patient morbidity.

III. Prospectively measure the effect of an automated notification program on adherence rates.

SECONDARY OBJECTIVES:

I. Quantify any time savings realized by patient care staff through the use of such a program.

II. Quantify the number of patient care interventions that directly result from this automated monitoring and notification program.

OUTLINE:

Patients' electronic medical records are reviewed for adherence, severe myelosuppression, and patient morbidity retrospectively and prospectively.

ELIGIBILITY:
Inclusion Criteria:

* RETROSPECTIVE: All patients seen in Dr. Lesser's clinic who received concurrent temozolomide and radiation therapy followed by adjuvant temozolomide for newly diagnosed malignant gliomas from 01/01/07 through 03/31/2010 will be analyzed
* PROSPECTIVE: All patients seen in Dr. Lesser's clinic who receive concurrent temozolomide and radiation therapy followed by adjuvant temozolomide for newly diagnosed malignant gliomas during and after the construction of the system until the end of the study

Exclusion Criteria:

* Patients participating in clinical trials or other deviations from non-standard therapies that engender similar monitoring risk will be evaluated for this study on a case by case basis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Brain Tumor Patients
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2015-02-23 (Actual); Study Completion 2015-02-23 (Actual)

PRIMARY OUTCOMES:
Frequency of nonadherence (retrospective) | Up to 42 days (completion of treatment)
  A two-sided 95.0% confidence interval for a single proportion using the large sample normal approximation will be extended from 8.1% in the observed proportion for an expected proportion of 25% non-adherence.
Impact of nonadherence events on myelosuppression severity (retrospective) | Up to 90 days after completion of treatment
  Severe myelosuppression will be defined as grade 3 or grade 4 myelosuppression from Common Terminology Criteria for Adverse Events version 3.0 criteria. The dates of any severe myelosuppressive events will be recorded. A Fisher's exact test with a 0.050 two-sided significance level will be used.
Impact of nonadherence events on patient morbidity (retrospective) | Up to 90 days after completion of treatment
  Patient morbidity (including date of event) will be assessed on all participants with severe myelosuppression, and includes: death during treatment with temozolomide or up to 90 days after treatment, the number of transfusions received for myelosuppression during treatment with temozolomide or up to 90 days after treatment, and the length of the hospital stay for myelosuppression during treatment with temozolomide or up to 90 days after treatment. A Fisher's exact test with a 0.050 two-sided significance level will be used.
Effect of an automated notification program on adherence rates (prospective) | Up to 6 years
  To compare the rates of adherence between the retrospective and prospective time periods, a Fisher's exact test with a 0.050 two-sided significance level will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Lesser, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States